CLINICAL TRIAL: NCT05391282
Title: A Study on Internal Carotid Artery Blood Flow Velocity Changes in Prone, Head Tilt and Trendelenberg Position in Infants: an Observational Study Using Transfontanel Ultrasound
Brief Title: Internal Carotid Artery Blood Flow in Infants With Prone Position
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical associate professor, Seoul National University Hospital
Other Study IDs: 2204-162-1320
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ultrasound assessment — Transfontanel ultrasound assessment before and after prone positioning

SUMMARY:
Little is known about how implementation of prone position contributes to general anesthesia-induced decrease in cerebral blood flow in infants. The investigators investigated this question in participants undergoing untethering, hypothesizing that cardiorespiratory changes during this procedure would reduce cerebral perfusion.

ELIGIBILITY:
Inclusion Criteria:

* pediatric neurosurgical patients receiving surgery under prone position

Exclusion Criteria:

* patients diagnosed as hydrocephalus
* premature closure of fontanelle
* patients diagnosed as patent ductus arteriosus or other congenital heart disease.

Max Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric neurosurgical patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05-23 (Estimated); Primary Completion 2023-12-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Changes of internal carotid artery blood flow velocity | from induction of anesthesia to end of operation, about 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided